CLINICAL TRIAL: NCT01089517
Title: A Phase 2, Randomized, Double-Masked, Controlled Trial to Establish the Safety and Efficacy of Intravitreous Injections of E10030 (Anti-PDGF Pegylated Aptamer) Given in Combination With Lucentis in Subjects With Neovascular Age-Related Macular Degeneration
Brief Title: A Safety and Efficacy Study of E10030 (Anti-PDGF Pegylated Aptamer) Plus Lucentis for Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPH1001
Record Dates: First submitted 2010-03-12; First posted 2010-03-18 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2017-04

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lucentis (Active Comparator)
  Interventions: Drug: Lucentis
- E10030 low dose plus Lucentis (Experimental)
  Interventions: Drug: E10030 plus Lucentis
- E10030 high dose plus Lucentis (Experimental)
  Interventions: Drug: E10030 plus Lucentis

INTERVENTIONS:
Drug: E10030 plus Lucentis — once a month intravitreal injection
  Arms: E10030 high dose plus Lucentis; E10030 low dose plus Lucentis
Drug: Lucentis — 10 mg/mL intravitreal injection monthly
  Arms: Lucentis

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of E10030 intravitreous injection when administered in combination with Lucentis® against a control of Lucentis® alone in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1:1 ratio to the following dose groups:

* E10030 0.3 mg/eye + Lucentis® 0. 5 mg/eye
* E10030 1.5 mg/eye + Lucentis® 0. 5 mg/eye
* E10030 sham + Lucentis® 0. 5 mg/eye

Subjects will be treated with active E10030 or sham E10030 in combination with Lucentis® at Day 0, Week 4, Week 8, Week 12, Week 16 and Week 20.

Primary Efficacy Endpoint:

The primary efficacy endpoint is mean change in visual acuity from baseline at the Week 24 visit

Safety Endpoints:

Safety endpoints include adverse events, vital signs, ophthalmic variables [visual acuity, intraocular pressure (IOP), ophthalmic examination, color fundus photography, fluorescein angiograms (FA), optical coherence tomography (OCT)], and laboratory variables.

Approximately 444 subjects will be randomized into one of the three treatment cohorts (approximately 148 patients per dose group).

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal choroidal neovascularization (CNV) due to AMD

Exclusion Criteria:

Any of the following underlying diseases including:

* Diabetes mellitus
* History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV - see Appendix 19.6), history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or coronary artery revascularization within 6 months, or ventricular tachyarrhythmias requiring ongoing treatment.
* Clinically significant impaired renal or hepatic function.
* Stroke (within 12 months of trial entry).
* Any major surgical procedure within one month of trial entry.
* Known serious allergies to the fluorescein dye used in angiography (mild allergy amenable to treatment is allowable), to the components of the ranibizumab (Lucentis) formulation, or to the components of the E10030 formulation

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Palmetto Retinal Center, West Columbia, South Carolina, United States

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 449 patients at approximately 69 centers in North America, South America, Europe and Israel.
Groups:
- Lucentis: Sham/Lucentis 0.5 mg
- E10030 0.3 mg/Lucentis 0.5 mg: E10030 0.3 mg/Lucentis 0.5 mg
- E10030 1.5 mg/Lucentis 0.5 mg: E10030 1.5 mg/Lucentis 0.5 mg
Period: Overall Study
Arm/Group | Lucentis | E10030 0.3 mg/Lucentis 0.5 mg | E10030 1.5 mg/Lucentis 0.5 mg
Started | 148 | 149 | 152
Completed | 144 | 144 | 147
Not Completed | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- E10030 Low Dose Plus Lucentis: E10030 0.3 mg/Lucentis 0.5 mg
- E10030 High Dose Plus Lucentis: E10030 1.5 mg/Lucentis 0.5 mg
- Total: Total of all reporting groups
Arm/Group | Lucentis | E10030 Low Dose Plus Lucentis | E10030 High Dose Plus Lucentis | Total
Number analyzed (Participants) | 148 | 149 | 152 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 11 | 29
  >=65 years | 140 | 139 | 141 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (7.98) | 77.6 (8.19) | 77.8 (8.36) | 77.8 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 90 | 92 | 275
  Male | 55 | 59 | 60 | 174
Region of Enrollment [Number; unit: participants]
  United States | 47 | 51 | 53 | 151
  Europe | 87 | 85 | 82 | 254
  Israel | 10 | 10 | 14 | 34
  South America | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity From Baseline at the Week 24 Visit
Description: The primary efficacy endpoint is the mean change in visual acuity from baseline at the Week 24 visit
Time Frame: 24 Weeks
Population: Intent to Treat Population (last observation carried forward)
Measure: Mean (Standard Error); unit: ETDRS Letters
Arm/Group | Lucentis | E10030 0.3 mg/Lucentis 0.5 mg | E10030 1.5 mg/Lucentis 0.5 mg
Number analyzed (Participants) | 147 | 147 | 151
ETDRS Letters | 6.5 (1.09) | 8.8 (1.09) | 10.6 (1.07)

2. Secondary Outcome: The Proportion of Subjects Gaining 15 or More ETDRS Letters From Baseline at the Week 24 Visit
Description: The proportion of subjects gaining 15 or more ETDRS letters from baseline at the Week 24 visit
Time Frame: 24 weeks
Population: Intent to Treat Population (last observation carried forward)
Measure: Number; unit: % subjects (i.e gaining >/=15 letters)
Arm/Group | Lucentis | E10030 0.3 mg/Lucentis 0.5 mg | E10030 1.5 mg/Lucentis 0.5 mg
Number analyzed (Participants) | 147 | 147 | 151
% subjects (i.e gaining >/=15 letters) | 34.0 | 33.3 | 39.1

3. Secondary Outcome: Proportion of Patients With at Least 1 Adverse Event
Time Frame: 24 weeks
Population: Safety Analysis Population
Measure: Number; unit: % of patients with adverse events
Arm/Group | Lucentis | E10030 0.3 mg/Lucentis 0.5 mg | E10030 1.5 mg/Lucentis 0.5 mg
Number analyzed (Participants) | 148 | 149 | 152
% of patients with adverse events | 65.5 | 67.1 | 65.1

ADVERSE EVENTS:
Arm/Group | Lucentis | E10030 Low Dose Plus Lucentis | E10030 High Dose Plus Lucentis
Serious Adverse Events (participants affected / at risk) | 12/148 | 14/149 | 10/152
Other Adverse Events (participants affected / at risk) | 63/148 | 63/149 | 69/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lucentis (N=148) | E10030 Low Dose Plus Lucentis (N=149) | E10030 High Dose Plus Lucentis (N=152)
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Corneal Erosion (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Rectal Hemmorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary Tract infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung squamous cell carcinoma, unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 2 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0
Vascular Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Mental status change (Psychiatric disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Arterial Disorder (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lucentis (N=148) | E10030 Low Dose Plus Lucentis (N=149) | E10030 High Dose Plus Lucentis (N=152)
Conjunctival hemorrhage (Eye disorders) | 37 | 34 | 51
Punctate Keratitis (Eye disorders) | 10 | 19 | 15
Eye Pain (Eye disorders) | 8 | 10 | 13
Conjunctival hyperemia (Eye disorders) | 13 | 9 | 13
Subretinal fibrosis (Eye disorders) | 8 | 6 | 5
Intraocular pressure increased (Investigations) | 4 | 8 | 9
Hypertension (Vascular disorders) | 8 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual site or investigator may publish or present any results from the trial until a joint, multi center publication of the trial results is made by Sponsor in conjunction with various participating investigators and appropriate sites contributing data and comments. Subsequently, individual investigators may request to publish or present results from the trial; however, approval will be at the sole discretion of the Sponsor.